CLINICAL TRIAL: NCT01322438
Title: A Phase 1, Non-Randomized, Open Label Study to Determine the Effect of Rifampin on the Pharmacokinetics of a Single Oral Dose of 160 mg Regorafenib (BAY73-4506) in Healthy Volunteers
Brief Title: Effect of Rifampin on the Pharmacokinetics of BAY73-4506
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15524
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Neoplasms
Keywords: healthy volunteers; rifampin; pharmacokinetics; single dose
MeSH Terms: conditions — Neoplasms | interventions — regorafenib; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Regorafenib (BAY73-4506) + rifampin

INTERVENTIONS:
Drug: Regorafenib (BAY73-4506) + rifampin — Drug: BAY73-4506 A single 160-mg dose of BAY73-4506 will be administered in the fasted state on Day 1 as four 40 mg tablets. Drug: BAY73-4506 and rifampin 600 mg once a day doses of rifampin will be orally administered after overnight fasting from Day 15 to Day 23. A single 160-mg dose of BAY73-4506 will be administered in the fasted state on Day 21 as four 40 mg tablets.

SUMMARY:
The purpose of this study is to see if giving rifampin, a marketed antibiotic, changes how your body absorbs and distributes BAY73-4506.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject
* Age: 18 to 45 years (inclusive) at the first screening examination / visit
* Body mass index (BMI): 18 to 32 kg/m² (inclusive)
* Ability to understand and follow study-related instructions
* Subjects enrolled in this study must use adequate barrier birth control measures prior to, during the course of the study, and 3 months after the last administration of regorafenib. An adequate contraception includes the use of condoms or a vasectomy. In addition, adequate birth control measures for the subject's partner is required, such as a hormonal contraception with implants or combined oral contraceptives, certain intrauterine devices, bilateral tubal ligation, or hysterectomy.

Exclusion Criteria:

* Clinically significant disease or condition
* Recent serious infection

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile | after 1 month
Proportion of subjects with adverse event collection | after 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Austin, Texas, United States